CLINICAL TRIAL: NCT03249454
Title: Effects of Transcutaneous Spinal Direct Current Stimulation in Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: TIRR/Mission Connect (Other)
Responsible Party: Principal Investigator, Radha Korupolu, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-17-0166
Record Dates: First submitted 2017-08-02; First posted 2017-08-15 (Actual); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-01

CONDITIONS: Incomplete Spinal Cord Injury
Keywords: Incomplete SCI

STUDY DESIGN:
Intervention Model Description: Crossover design with 9 arms: Anodal tsDCS, Cathodal tsDCS, Sham tsDCS
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (11):
- Anode, then Cathode, then Anode, then Sham, then Cathode tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS
- Sham, then Cathode, then Anode, then Anode, then Cathode tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS
- Anode, then Cathode, then Sham, then Anode, then Cathode tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS
- Cathode, then Anode, then Cathode, then Anode, then Sham tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS
- Anode, then Anode, then Sham, then Cathode, then Cathode tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS
- Sham, then Anode, then Cathode, then Cathode, then Anode tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS
- Cathode, then Anode, then Cathode, then Sham, then Anode tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS
- Sham, then Anode, then Cathode, then Anode, then Cathode tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS
- Cathode, then Cathode, then Sham, then Anode, then Anode tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS
- Anode, Then Cathode, Then Anode, Then Cathode Then Sham tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS
- Sham, Then Anode, Then Anode, Then Cathode, Then Cathode tsDCS (Experimental): 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
  Interventions: Device: Anodal tsDCS; Device: Cathodal tsDCS; Device: Sham tsDCS

INTERVENTIONS:
Device: Anodal tsDCS — During Anodal tsDCS intervention the positive end of the battery will be connected to the electrode on participant's back and negative end of the battery will be connected to the electrode on participant's shoulder. The battery will be turned on for 15 minutes, and the stimulation strength will be adjusted a couple of times per tolerance level.
Device: Cathodal tsDCS — During Cathodal tsDCS intervention the negative end of the battery will be connected to the electrode on participant's back and positive end of the battery will be connected to the electrode on participant's shoulder. The battery will be turned on for 15 minutes, and the stimulation strength will be adjusted a couple of times per tolerance level.
Device: Sham tsDCS — During Sham tsDCS intervention, battery will be turned off and no current will pass through the electrodes.

SUMMARY:
The purpose of the study is to investigate the effects of a novel therapeutic approach with transcutaneous spinal direct current stimulation (tsDCS) to promote functional recovery and spasticity in chronic spinal cord injury (SCI).

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effects of a novel therapeutic approach to promote functional recovery and spasticity in chronic SCI. The tsDCS effect on neuro-physiological measures such as H reflex and somatosensory evoked potential (SSEP) wiil be evaluated in subjects with SCI. This incremental, design will allow the establishment of strong electrophysiological data prior to rapid clinical translation of the findings about this promising, early-stage technique.

The central hypothesis is twofold: 1) active tsDCS will lead to a change in Hmax/M max ratio than sham tsDCS, in a polarity dependent manner; and 2) active tsDCS will lead to a change in SSEP amplitude and latency, in a polarity dependent manner.

ELIGIBILITY:
Inclusion Criteria:

* Providing written informed consent prior to any study related procedures
* 18-65 years of age
* Motor incomplete SCI classified as B, C or D by the American Spinal Injury Association Impairment Scale (AIS)
* Traumatic lesion at or above T8-T9 neurological level
* Body mass index ≤ 30 (in order to facilitate reliable location of body landmarks guiding stimulation);
* Chronic SCI (time since injury>6 months)

Exclusion Criteria:

* Unstable cardiopulmonary conditions
* History of seizure, head injury with loss of consciousness, severe alcohol or drug abuse, and/or psychiatric illness
* Any joint contracture or severe spasticity, as measured by a Modified Ashworth Score 4
* Subject who cannot provide self-transportation to the study location
* Cardiac or neural pacemakers
* Pregnancy
* lower motor neuron injury (eg: peripheral neuropathy, cauda equina syndrome)
* Uncontrolled diabetes with HbA1C>7
* History of severe autonomic dysreflexia
* No planned alteration in therapy or medication for muscle tone during the course of the study(No botulinum toxin injections in last 3 months, No phenol injections in last 6 months, intrathecal baclofen pump dose stable for past 3 months, etc)
* Conditions for e.g., severe arthritis, extreme shoulder pain that would interfere with valid administration of the measures or with interpreting motor testing;
* No contraindications to tsDCS
* ferromagnetic material in the brain or in the spine (except for titanium used in segmental)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Radha Korupolu, MD, Principal Investigator — The University of Texas Health Science Center
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 15 subjects.
Pre-assignment Details: 2 enrolled participants were not assigned to an arm--one of these participant had leg edema that interfered with outcome assessment, and the second participant did not exhibit an H reflex due to a baclofen medication pump; therefore, these 2 participants were not randomized and did not start any intervention.
Groups:
- Anode, Then Cathode, Then Anode, Then Sham, Then Cathode tsDCS: 5 transcutaneous spinal direct current stimulation (tsDCS) sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
Period: Overall Study
Arm/Group | Anode, Then Cathode, Then Anode, Then Sham, Then Cathode tsDCS | Sham, Then Cathode, Then Anode, Then Anode, Then Cathode tsDCS | Anode, Then Cathode, Then Sham, Then Anode, Then Cathode tsDCS | Cathode, Then Anode, Then Cathode, Then Anode, Then Sham tsDCS | Anode, Then Anode, Then Sham, Then Cathode, Then Cathode tsDCS | Sham, Then Anode, Then Cathode, Then Cathode, Then Anode tsDCS | Cathode, Then Anode, Then Cathode, Then Sham, Then Anode tsDCS | Sham, Then Anode, Then Cathode, Then Anode, Then Cathode tsDCS | Cathode, Then Cathode, Then Sham, Then Anode, Then Anode tsDCS | Anode, Then Cathode, Then Anode, Then Cathode Then Sham tsDCS | Sham, Then Anode, Then Anode, Then Cathode, Then Cathode tsDCS
Started | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1
First Intervention (1 Day) | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Washout (1 Week) | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Second Intervention (1 Day) | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Washout (1 Week) | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Third Intervention (1 Day) | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Washout (1 Week) | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Fourth Intervention (1 Day) | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Washout (1 Week) | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Fifth Intervention (1 Day) | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Completed | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: 5 tsDCS sessions were performed for each subject, with at least a 1 week washout period between tsDCS sessions. For each session, the subject was randomly assigned to cathodal, anodal or sham tsDCS. Each subject who completed the study received 2 cathodal, 2 anodal and 1 sham tsDCS session.
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.40 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 4
  Asian | 1
  Caucasian | 7
  Hispanic/Latino | 2
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Height [Mean (Standard Deviation); unit: centimeters] | 173.05 (7.90)
Weight [Mean (Standard Deviation); unit: kilograms] | 76.69 (16.92)
Employment Status [Count of Participants; unit: Participants]
  Employed | 3
  Unemployed | 11
  Student | 1
Marital Status [Count of Participants; unit: Participants]
  Single | 7
  Engaged | 1
  Married | 5
  Divorced | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Hmax
Description: Immediately before application of tsDCS and after application of tsDCS, Hmax will be obtained from soleus muscle by stimulation of tibial nerve. The H-reflex is a compound muscle action potential elicited by low-threshold electrical stimulation of afferent fibers in the mixed nerve with subsequent monosynaptic excitation of alpha motoneurons. Changes in the excitability of the reflex pathway are estimated by measuring the amplitude of the reflex.
Time Frame: 10 minutes before intervention, 10 minutes after intervention
Population: Those who completed the study were analyzed. Data are reported per session. There were potentially 22 cathode, 22 anode, and 11 sham sessions. Data for the Right Lower Extremity were not collected for 3 cathode, 3 anode, and 2 sham sessions, and data for the Left Lower Extremity were not collected for 3 cathode, 1 anode, and 2 sham sessions.
Measure: Mean (Standard Deviation); unit: percent change in Hmax
Units Other Than Participants: sessions
Groups:
- Cathodal tsDCS: Each subject will be assigned to receive two cathodal tsDCS interventions randomly. There will be at least 1 week washout period between any 2 sessions.
  Cathodal tsDCS: During Cathodal tsDCS intervention the negative end of the battery will be connected to the electrode on participant's back and positive end of the battery will be connected to the electrode on participant's shoulder. The battery will be turned on for 15 minutes, and the stimulation strength will be adjusted a couple of times per tolerance level.
- Anodal tsDCS: Each subject will be assigned to receive two anodal tsDCS interventions randomly. There will be at least 1 week washout period between any 2 sessions.
  Anodal tsDCS: During Anodal tsDCS intervention the positive end of the battery will be connected to the electrode on participant's back and negative end of the battery will be connected to the electrode on participant's shoulder. The battery will be turned on for 15 minutes, and the stimulation strength will be adjusted a couple of times per tolerance level.
- Sham tsDCS: Each subject will be assigned to receive one sham tsDCS interventions randomly. There will be at least 1 week washout period between any 2 sessions.
  Sham tsDCS: During Sham tsDCS intervention, battery will be turned off and no current will pass through the electrodes.
Arm/Group | Cathodal tsDCS | Anodal tsDCS | Sham tsDCS
Number analyzed (Participants) | 11 | 11 | 11
Number analyzed (sessions) | 19 | 21 | 9
percent change in Hmax
  Right Lower Extremity: number analyzed (Participants) | 10 | 10 | 9
  Right Lower Extremity: number analyzed (sessions) | 19 | 19 | 9
  Right Lower Extremity | 27.85 (63.57) | 8.43 (29.21) | -4.91 (39.12)
  Left Lower Extremity | 16.20 (55.37) | -3.99 (23.04) | 34.04 (94.72)

2. Primary Outcome: Change in Somatosensory Evoked Potential (SSEP)
Description: A somatosensory evoked potential (SSEP) is the electrical activity response measured at the skin's surface along ascending sensory pathway following controlled peripheral nerve stimulation by tsDCS. For recording posterior tibial nerve SSEPs, the nerve is stimulated at the ankle, with the cathode midway between the Achilles tendon and the medial malleolus and the anode 3 cm distal to the cathode. Nerve stimulation should consist of a 0.1-0.2 ms duration square wave pulse at 3-5 Hertz (Hz). These pulses will be delivered by constant voltage stimulator applied transcutaneously over the targeted nerve. The stimulation intensity would exceed the motor threshold for eliciting a muscle twitch. Electromyogram (EMG)/ Nerve Conduction Velocity (NCV) measuring system will be used to measure SSEPs.
Time Frame: 30 to 40 minutes before intervention, 30 to 40 minutes after intervention
Population: Data was not collected for this outcome measure.
Arm/Group | Cathodal tsDCS | Anodal tsDCS | Sham tsDCS
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change Systolic Blood Pressure
Description: Systolic Blood pressure will be recorded before and after each tsDCS session.
Time Frame: 60 to 90 minutes before intervention, 60 to 90 minutes after intervention
Population: Those who completed the study were analyzed. Data are reported per session. After randomization, there were potentially 22 cathode sessions, 22 anode sessions, and 11 sham sessions--of these sessions, data were not collected for 2 cathode sessions, 3 anode sessions, and 2 sham sessions.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Units Other Than Participants: sessions
Arm/Group | Cathodal tsDCS | Anodal tsDCS | Sham tsDCS
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (sessions) | 20 | 19 | 9
millimeters of mercury (mmHg) | 7.90 (13.31) | 7.58 (10.37) | -4.00 (6.68)

4. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Diastolic Blood pressure will be recorded before and after delivering each intervention
Time Frame: 60 to 90 minutes before intervention,60 to 90 minutes after intervention ( for each intervention)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Units Other Than Participants: sessions
Arm/Group | Cathodal tsDCS | Anodal tsDCS | Sham tsDCS
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (sessions) | 20 | 19 | 9
millimeters of mercury (mmHg) | 4.80 (15.07) | 2.16 (6.65) | -0.44 (9.06)

5. Secondary Outcome: Change in Heart Rate
Description: Heart rate will be recorded before and after delivering each intervention
Time Frame: 60 to 90 minutes before intervention,60 to 90 minutes after intervention ( for each intervention)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Units Other Than Participants: sessions
Arm/Group | Cathodal tsDCS | Anodal tsDCS | Sham tsDCS
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (sessions) | 20 | 19 | 9
beats per minute (bpm) | -7.35 (5.28) | -6.53 (6.99) | -4.78 (5.63)

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: The urinary tract infection (UTI) was unrelated to the intervention--this subject developed a UTI after randomization and completion of one anodal stimulation session.
  Bruising was related to outcome measure collection (that is, related to preparation for measurement of h-reflex, which involves cleaning of the skin and placing electrodes) but unrelated to the intervention--this subject withdrew after randomization and completion of one session of sham stimulation.
Arm/Group | Cathodal tsDCS | Anodal tsDCS | Sham tsDCS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cathodal tsDCS (N=15) | Anodal tsDCS (N=15) | Sham tsDCS (N=15)
Hospitalization for Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cathodal tsDCS (N=15) | Anodal tsDCS (N=15) | Sham tsDCS (N=15)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size. We did not control for timing of oral anti-spasticity medications during different trials which can effect H reflex measurement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03249454/Prot_SAP_000.pdf